CLINICAL TRIAL: NCT00168428
Title: A Study Using Botulinum Toxin Type A as Headache Prophylaxis for Migraine Patients With Frequent Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-080
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-10

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- botulinum toxin Type A (Experimental): Two treatment sessions in the double-blind phase and three treatment sessions in the open-label extension phase. Total minimum dose is 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas with the total maximum dose of 195 U with 39 head/neck injections.
  Interventions: Biological: Botulinum Toxin Type A
- Placebo (saline) (Placebo Comparator): Two treatment sessions in the double-blind phase. Total minimum dose in 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas and the total maximum dose is 195 U with 39 head/neck injections.
  Interventions: Other: placebo (saline)

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Two treatment sessions in the double-blind phase and three treatment sessions in the open-label phase. Total minimum dose is 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas with the total maximum dose of 195 U with 39 head/neck injections.
  Other Names: BOTOX®
  Arms: botulinum toxin Type A
Other: placebo (saline) — Two treatment sessions in the double-blind phase. Total minimum dose in 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas and the total maximum dose is 195 U with 39 head/neck injections.
  Arms: Placebo (saline)

SUMMARY:
This is a 60 week study including a double-blind phase followed by an open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Frequent migraine (>=15 headache days per month)
* >=4 distinct headache episodes lasting >=4 hours
* >=50% of baseline headache days migraine/probable migraine days

Exclusion Criteria:

* Previous use of botulinum toxin of any serotype or immunization to any botulinum toxin serotype
* Any medical condition that puts the patient at increased risk with exposure to BOTOX
* Diagnosis of complicated migraine, chronic tension-type headache, hypnic headache, hemicrania continua, new daily persistent headache
* Use of prophylactic headache medication within 28 days prior to week -4
* Unremitting headache lasting continuously throughout the 4-week baseline period
* Known or suspected TMD
* Diagnosis of fibromyalgia
* Beck depression inventory score >24 at week-4
* Psychiatric problems that may have interfered with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Walnut Creek, California, United States
- Calgary, Alberta, Canada
- Zagreb, Croatia
- Essen, Germany
- Zurich, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Diener HC, Dodick DW, Lipton RB, Manack Adams A, DeGryse RE, Silberstein SD. Benefits Beyond Headache Days With OnabotulinumtoxinA Treatment: A Pooled PREEMPT Analysis. Pain Ther. 2020 Dec;9(2):683-694. doi: 10.1007/s40122-020-00198-w. Epub 2020 Oct 7. PMID 33026631
- [Derived] Silberstein SD, Diener HC, Dodick DW, Manack Adams A, DeGryse RE, Lipton RB. The Impact of OnabotulinumtoxinA vs. Placebo on Efficacy Outcomes in Headache Day Responder and Nonresponder Patients with Chronic Migraine. Pain Ther. 2020 Dec;9(2):695-707. doi: 10.1007/s40122-020-00199-9. Epub 2020 Oct 7. PMID 33026630
- [Derived] Dodick DW, Silberstein SD, Lipton RB, DeGryse RE, Adams AM, Diener HC. Early onset of effect of onabotulinumtoxinA for chronic migraine treatment: Analysis of PREEMPT data. Cephalalgia. 2019 Jul;39(8):945-956. doi: 10.1177/0333102418825382. Epub 2019 May 21. PMID 31112399
- [Derived] Silberstein SD, Dodick DW, Aurora SK, Diener HC, DeGryse RE, Lipton RB, Turkel CC. Per cent of patients with chronic migraine who responded per onabotulinumtoxinA treatment cycle: PREEMPT. J Neurol Neurosurg Psychiatry. 2015 Sep;86(9):996-1001. doi: 10.1136/jnnp-2013-307149. Epub 2014 Dec 12. PMID 25500317
- [Derived] Rendas-Baum R, Yang M, Varon SF, Bloudek LM, DeGryse RE, Kosinski M. Validation of the Headache Impact Test (HIT-6) in patients with chronic migraine. Health Qual Life Outcomes. 2014 Aug 1;12:117. doi: 10.1186/s12955-014-0117-0. PMID 25080874
- [Derived] Aurora SK, Winner P, Freeman MC, Spierings EL, Heiring JO, DeGryse RE, VanDenburgh AM, Nolan ME, Turkel CC. OnabotulinumtoxinA for treatment of chronic migraine: pooled analyses of the 56-week PREEMPT clinical program. Headache. 2011 Oct;51(9):1358-73. doi: 10.1111/j.1526-4610.2011.01990.x. Epub 2011 Aug 29. PMID 21883197
- [Derived] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038

RESULTS

PARTICIPANT FLOW:
Period: Double-Blind Phase (DB)
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Started | 347 | 358
Completed | 311 (Completed Week 24) | 334 (Completed Week 24)
Not Completed | 36 | 24
Period: Open-Label Phase (OL)
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Started | 305 (Number of DB Botulinum toxin type A patients who rolled into OL phase) | 329 (Number of DB Placebo patients who rolled into OL phase)
Completed | 261 | 261
Not Completed | 44 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo (Saline) | Total
Number analyzed (Participants) | 347 | 358 | 705
Age, Customized [Number; unit: participants]
  < 40 years | 149 | 160 | 309
  >= 40 years | 198 | 198 | 396
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 303 | 602
  Male | 48 | 55 | 103

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Headache Days
Description: Mean change from baseline in frequency (number) of headache days during the 28 day period ending with Week 24. Headache day defined as a calendar day [00:00 to 23:59] for which the patient reported >= 4 continuous hours of headache.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Headache Days
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Headache Days
  Baseline | 19.9 (3.63) | 19.7 (3.65)
  Change from Baseline at Week 24 | -9.0 (6.54) | -6.7 (6.67)

2. Secondary Outcome: Change in Total Cumulative Hours of Headache Occurring on Headache Days
Description: Mean change from baseline in total cumulative hours of headache occurring on headache days during the 28 day period ending with Week 24. Headache day defined as a calendar day [00:00 to 23:59] when the patient reported >= 4 continuous hours of headache.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Hours
  Baseline | 296.18 (121.043) | 287.20 (118.089)
  Change from Baseline at Week 24 | -132.41 (130.216) | -90.01 (133.758)

3. Secondary Outcome: Change in Frequency of Moderate/Severe Headache Days
Description: Mean change from baseline in frequency (number) of moderate/severe headache days during the 28 day period ending with Week 24. Those calendar days with >= 4 continuous hours of headache were selected. As per the patient diary, all headache episodes occurring during those days with a maximum severity of moderate or severe were counted.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Moderate/Severe Headache Days
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Moderate/Severe Headache Days
  Baseline | 18.1 (4.03) | 17.7 (4.26)
  Change from Baseline at Week 24 | -8.3 (6.37) | -5.8 (6.59)

4. Secondary Outcome: Change in Frequency of Migraine/Probable Migraine Headache Days
Description: Mean change from baseline in frequency (number) of migraine/probable migraine headache days during the 28 day period ending with Week 24. Headache day defined as a calendar day with >= 4 continuous hours of headache meeting the ICHD-II criteria for migraine or probable migraine.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Migraine/Probable Migraine Headache Days
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Migraine/Probable Migraine Headache Days
  Baseline | 19.2 (3.94) | 18.7 (4.05)
  Change from Baseline at Week 24 | -8.7 (6.64) | -6.3 (6.71)

5. Secondary Outcome: Change in Frequency of Headache Episodes
Description: Mean change from baseline in frequency (number) of headache episodes during the 28 day period ending with Week 24. Headache episode defined as patient-reported headache with a start and stop time indicating that the pain lasted >= 4 continuous hours.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Headache Episodes
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Headache Episodes
  Baseline | 12.0 (5.27) | 12.7 (5.29)
  Change from Baseline at Week 24 | -5.3 (5.12) | -4.6 (4.84)

6. Secondary Outcome: Percentage of Patients With Severe HIT-6 Impact Category Scores
Description: Percentage of patients with a severe (60-78) score on the Headache Impact Test (HIT-6) Questionnaire during the 28 day period, ending with Week 24. The HIT-6 consisted of 6 questions about headache and impact on the patient's health and well-being. Answers for each question ranged from 6=Never, 8=Rarely, 10=Sometimes, 11=Very Often, and 13=Always. The total scores ranged from 36-49 (Little or No Impact), 50-55 (Some Impact), 56-59 (Substantial Impact) and 60-78 (Severe Impact).
Time Frame: Week 24
Population: Intent to Treat
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 347 | 358
Percentage of Patients | 66.3 | 76.5

ADVERSE EVENTS:
Description: For SAEs/AEs, the Total # Participants at Risk for the Botulinum toxin type A arm includes ALL patients in the safety population who received Botulinum toxin type A in the Double-Blind and Open-Label phases. The total # Participants at Risk for the Placebo arm includes ONLY Double-blind Phase patients in the safety population who received Placebo.
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Serious Adverse Events (participants affected / at risk) | 33/676 | 8/358
Other Adverse Events (participants affected / at risk) | 195/676 | 34/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=676) | Placebo (Saline) (N=358)
Migraine (Nervous system disorders) | 4 | 1
Pneumonia (Infections and infestations) | 3 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=676) | Placebo (Saline) (N=358)
Neck pain (Musculoskeletal and connective tissue disorders) | 61 | 8
Nasopharyngitis (Infections and infestations) | 47 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 47 | 2
Sinusitis (Infections and infestations) | 40 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.